CLINICAL TRIAL: NCT05151224
Title: Circulating microRNA 21 Expression Level Before and After Neoadjuvant Systemic Therapy in Breast Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ebtehal Mohamed Mahmoud Salah, Dr., Ain Shams University
Other Study IDs: FMASUMD232/2021
Record Dates: First submitted 2021-11-27; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Breast Carcinoma
Keywords: breast, microRNA 21, Neoadjuvant thera[py
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients eligible to neoadjuvant systemic therapy: Invasive breast cancer, age are 18 years or more, from stage IIB to stage IIIC, all subtypes are included, either HR (ER, PR) positive or negative, HER2 positive or negative, eligible to neoadjuvant systemic therapy.
  Interventions: Diagnostic Test: microRNA 21

INTERVENTIONS:
Diagnostic Test: microRNA 21 — Plasma microRNA 21 5p expression, by real-time polymerase chain reaction, before and after neoadjuvant systemic therapy.
  Blood sample will be taken by a trained nurse, amount of blood will be 3 ml, and will be taken twice, one time before the start of the neoadjuvant systemic treatment , second time by the end of the neoadjuvant systemic treatment.

SUMMARY:
MicroRNAs (miRNAs) are involved in the development and progression of malignant tumors. In breast cancer, differential miRNA expression has been demonstrated across breast cancer subtypes, with both tumor-promoting and tumor suppressive functions for individual miRNAs.

Novel predictive biomarkers that can be assessed in the liquid specimen before systemic treatment could help to individualize treatment decisions in breast cancer and to potentially avoid ineffective systemic treatment.

In our study we detect level of circulating miRNA 21 in breast cancer patient before and after neoadjuvant treatment , whether there will be change or not, and if related to complete pathological response.

DETAILED DESCRIPTION:
MicroRNAs (miRNAs) are a group of non-coding, single stranded RNAs of ~ 19-24 nucleotides, which act by a novel mechanism of posttranscriptional regulation that is profoundly altered in malignant cells. (Ling, Fabbri and Calin, 2013).Based on the function of miRNAs, they are divided into two types: an oncomir, implicated in cancer progression by regulating tumor suppressor genes negatively; and a tumor suppressor, preventing cancers by regulating oncogenes. (Zhang et al., 2007).

A key oncomir in carcinogenesis is miRNA-21, which was one of the first miRNAs detected in the human genome. It is located on chromosome 17 in the tenth intron of the coding gene transmembrane protein 49, which targets various tumor suppressors like PTEN, PDCD4, p53, and TAp63 pathways. (Yadav et al., 2016)

Experimental and literature research has highlighted that miRNA-21 was always significantly elevated in every study that included invasive breast carcinomas compared with healthy breast tissue. (Petrović, 2016).

miRNA-21 has been shown to be a very important promoter of cellular outgrowth, migration, invasion, and metastasis. In breast carcinoma cell lines, miRNA-21 was connected to cell proliferation and migration. (Yan et al., 2011).

Mei and her colleagues (2010) reported that miRNA-21 up-regulation is associated with therapy (taxol) resistance in breast cancer cells and further validated in a recent study by (Chen and Bourguignon, 2014) in which miRNA-21 up-regulation resulted in an increase of anti-apoptosis protein BCL-2 and chemo-resistance in breast cancer cells

Various studies have supported the potential role of circulating miRNAs to be used as prognostic and predictor biomarkers in breast cancer. (Schwarzenbach, 2017)

In their analysis of the blood serum of 56 breast cancer patients, Wang et al. (2012) illustrate reduced miR-125b levels to correlate with resistance to four cycles of neoadjuvant 5-fluorouracil, epirubicin and cyclophosphamide (FEC). Another recent study investigating dynamic changes of circulating miRNA as indicator for clinical response for neoadjuvant chemotherapy in HER2 negative patients , found that dynamics of three plasma miRNA , including miRNA 222, miRNA 20-a and miRNA 451 was associated with chemosensitivity. (Zhu et al., 2018)

The expression of serum-miRNA-125b and the changes of serum miRNA-21 expression during neoadjuvant chemotherapy were associated with chemotherapy response and disease-free survival (DFS). (Liu et al., 2017). Yadav et al. (2016) found that breast cancer patients received neoadjuvant therapy shows significant impact on overall reduction in serum miRNA-21 expression compared to before therapy (p < 0.0001)

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years old.
* Breast cancer diagnosis histologically proven and pathology report from breast and ipsilateral axillary nodes.
* Pathology: invasive carcinoma.
* Staging: tumor size >2cm (>/=T2), node positive (N >/= 1), i.e. >/= T2N1; from stage IIB to stage IIIC, according to AJCC breast Cancer staging 8th edition. (Giuliano, Edge and Hortobagyi, 2018)
* All subtypes are included, either HR (ER, PR) positive or negative, HER2 positive or negative.
* Neoadjuvant systemic treatment composed of anthracyclines-based chemotherapy and taxanes, trastuzumab for HER2 positive patients

Exclusion Criteria:

* Metastatic breast cancer
* inflammatory breast cancer,
* male breast cancer,
* bilateral breast cancer, or concurrent malignancy
* Previous malignancy.
* Presence of any contraindication to neoadjuvant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasive breast cancer, from stage IIB to stage IIIC, all subtypes are included, who are candidates for neoadjuvant systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Describe miRNA 21 expression level before and after neoadjuvant systemic therapy in breast cancer patient. | 1 year
  miRNA 21 expression level before and after neoadjuvant systemic therapy

SECONDARY OUTCOMES:
Measure relation between miRNA 21 expression level before and after neoadjuvant systemic therapy and pathological response. | 1 year
  Relation between miRNA 21 expression level before and after neoadjuvant systemic therapy and pathological response
Measure relation between the miRNA 21 expression and the clinicopathological parameters of Breast Cancer patients. | 1 year
  Relation between the miRNA 21 expression and the clinicopathological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ebtehal M Salah, Principal Investigator — Assistant lecturer of clinical oncology; Iman Sharawy, Study Director — Professor of clinical oncology
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mei M, Ren Y, Zhou X, Yuan XB, Han L, Wang GX, Jia Z, Pu PY, Kang CS, Yao Z. Downregulation of miR-21 enhances chemotherapeutic effect of taxol in breast carcinoma cells. Technol Cancer Res Treat. 2010 Feb;9(1):77-86. doi: 10.1177/153303461000900109. PMID 20082533
- [Result] Yadav P, Mirza M, Nandi K, Jain SK, Kaza RC, Khurana N, Ray PC, Saxena A. Serum microRNA-21 expression as a prognostic and therapeutic biomarker for breast cancer patients. Tumour Biol. 2016 Nov;37(11):15275-15282. doi: 10.1007/s13277-016-5361-y. Epub 2016 Sep 30. PMID 27696295
- [Result] Ling H, Fabbri M, Calin GA. MicroRNAs and other non-coding RNAs as targets for anticancer drug development. Nat Rev Drug Discov. 2013 Nov;12(11):847-65. doi: 10.1038/nrd4140. PMID 24172333
- [Result] Zhang B, Pan X, Cobb GP, Anderson TA. microRNAs as oncogenes and tumor suppressors. Dev Biol. 2007 Feb 1;302(1):1-12. doi: 10.1016/j.ydbio.2006.08.028. Epub 2006 Aug 16. PMID 16989803
- [Result] Petrovic N. miR-21 Might be Involved in Breast Cancer Promotion and Invasion Rather than in Initial Events of Breast Cancer Development. Mol Diagn Ther. 2016 Apr;20(2):97-110. doi: 10.1007/s40291-016-0186-3. PMID 26891730
- [Result] Yan LX, Wu QN, Zhang Y, Li YY, Liao DZ, Hou JH, Fu J, Zeng MS, Yun JP, Wu QL, Zeng YX, Shao JY. Knockdown of miR-21 in human breast cancer cell lines inhibits proliferation, in vitro migration and in vivo tumor growth. Breast Cancer Res. 2011 Jan 10;13(1):R2. doi: 10.1186/bcr2803. PMID 21219636
- [Result] Chen L, Bourguignon LY. Hyaluronan-CD44 interaction promotes c-Jun signaling and miRNA21 expression leading to Bcl-2 expression and chemoresistance in breast cancer cells. Mol Cancer. 2014 Mar 8;13:52. doi: 10.1186/1476-4598-13-52. PMID 24606718
- [Result] Schwarzenbach H. Clinical Relevance of Circulating, Cell-Free and Exosomal microRNAs in Plasma and Serum of Breast Cancer Patients. Oncol Res Treat. 2017;40(7-8):423-429. doi: 10.1159/000478019. Epub 2017 Jun 28. PMID 28683441
- [Result] Zhu W, Liu M, Fan Y, Ma F, Xu N, Xu B. Dynamics of circulating microRNAs as a novel indicator of clinical response to neoadjuvant chemotherapy in breast cancer. Cancer Med. 2018 Sep;7(9):4420-4433. doi: 10.1002/cam4.1723. Epub 2018 Aug 11. PMID 30099860
- [Result] Wang H, Tan G, Dong L, Cheng L, Li K, Wang Z, Luo H. Circulating MiR-125b as a marker predicting chemoresistance in breast cancer. PLoS One. 2012;7(4):e34210. doi: 10.1371/journal.pone.0034210. Epub 2012 Apr 16. PMID 22523546
- [Result] Liu B, Su F, Chen M, Li Y, Qi X, Xiao J, Li X, Liu X, Liang W, Zhang Y, Zhang J. Serum miR-21 and miR-125b as markers predicting neoadjuvant chemotherapy response and prognosis in stage II/III breast cancer. Hum Pathol. 2017 Jun;64:44-52. doi: 10.1016/j.humpath.2017.03.016. Epub 2017 Apr 12. PMID 28412211